CLINICAL TRIAL: NCT00887471
Title: Comparison of Polysomnography Outcomes for Microdebrider-assisted Partial Intracapsular Tonsillectomy Versus Total Tonsillectomy
Brief Title: Comparison of Sleep Study Results After Partial Intracapsular Tonsillectomy Versus Total Tonsillectomy
Status: Completed | Type: Observational
Sponsor: State University of New York - Downstate Medical Center (Other)
Collaborators: American Society of Pediatric Otolaryngology (Other)
Responsible Party: Sponsor
Other Study IDs: 06-095
Record Dates: First submitted 2008-03-28; First posted 2009-04-24 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2012-06

CONDITIONS: Sleep-disordered Breathing; Obstructive Sleep Apnea
Keywords: Sleep-disordered breathing; Obstructive sleep apnea; Polysomnography; Tonsillectomy; Microdebrider assisted partial intracapsular tonsillectomy
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Adenoidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children who underwent PITA: Children who underwent partial intracapsular tonsillectomy and adenoidectomy between July 2003 and January 2008 for treatment of pediatric sleep-disordered breathing documented by positive preoperative polysomnography.
  Interventions: Procedure: PITA or T&A
- Children who underwent T&A: Children who underwent total tonsillectomy and adenoidectomy between July 2003 and January 2008 for treatment of pediatric sleep-disordered breathing documented by positive preoperative polysomnography.
  Interventions: Procedure: PITA or T&A

INTERVENTIONS:
Procedure: PITA or T&A — PITA - Microdebrider-assisted Partial Intracapsular Tonsillectomy and Adenoidectomy T&A - Bove Electrocautery Complete Tonsillectomy and Adenoidectomy
  Other Names: PITA = Partial Intracapsular Tonsillectomy and Adenoidectomy; T&A = Tonsillectomy and Adenoidectomy

SUMMARY:
The purpose of this study is to demonstrate similar improvements in sleep-disordered breathing as determined by sleep study with microdebrider-assisted partial intracapsular tonsillectomy and adenoidectomy versus total Bovie electrocautery tonsillectomy and adenoidectomy.

DETAILED DESCRIPTION:
Objectives: To demonstrate similar improvement in sleep-disordered breathing as determined by polysomnography (PSG) with microdebrider-assisted partial intracapsular tonsillectomy and adenoidectomy (PITA) versus Bovie electrocautery complete tonsillectomy and adenoidectomy (T&A).

Methods: In a retrospective cohort study children found to have Obstructive Sleep Apnea (OSA) by PSG who have undergone either PITA or T&A as treatment will be evaluated with repeat PSG. The groups will be matched by age, sex, and severity of pre-operative Apnea-Hypopnea Indices (AHI). The investigators performing and evaluating the PSG will be blinded to type of procedure and preoperative AHI. Change scores will be computed for each participant and the change scores of the groups compared.

ELIGIBILITY:
Inclusion Criteria:

* The medical records of 149 children who underwent partial intracapsular tonsillectomy and adenoidectomy at the State University of New York (SUNY) Downstate Medical Center or the Long Island College Hospital will be reviewed to identify children with positive preoperative polysomnography. 18 of those with positive preoperative studies will be randomly selected and offered participation in the study.
* Once enrolled, the participants will be matched by age, sex, time since procedure and polysomnography results (Apnea Hypopnea Index Index within 5) to 18 children who underwent traditional tonsillectomy and adenoidectomy (out of a total of 455 patients).

Exclusion Criteria:

* Recurrent tonsillitis
* Craniofacial syndromes
* Neuromuscular disorders
* Sickle cell disease

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children treated at the SUNY Downstate Medical Center or the Long Island College Hospital in Brooklyn, NY for sleep-disordered breathing documented by positive polysomnography by either Partial Intracapsular Tonsillectomy and Adenoidectomy or complete Tonsillectomy and Adenoidectomy between 2003 and 2008.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nira A Goldstein, MD, Principal Investigator — State University of New York - Downstate Medical Center; Jason R Mangiardi, MD, Study Director — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Result] Mangiardi J, Graw-Panzer KD, Weedon J, Regis T, Lee H, Goldstein NA. Polysomnography outcomes for partial intracapsular versus total tonsillectomy. Int J Pediatr Otorhinolaryngol. 2010 Dec;74(12):1361-6. doi: 10.1016/j.ijporl.2010.09.003. Epub 2010 Sep 28. PMID 20880595

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Review of surgical case logs identified 45 patients with positive polysomnography (PSG) (laboratory-based, home or nap)who had undergone PITA and 101 with positive PSG who had undergone T&A.
Pre-assignment Details: Of these 15 PITA patients entered and completed the study and 15 matched T&A patients entered and completed the study.
Groups:
- Children Who Underwent PITA: Children who underwent partial intracapsular tonsillectomy and adenoidectomy.
- Children Who Underwent T&A: Children who underwent total tonsillectomy and adenoidectomy.
Period: Overall Study
Arm/Group | Children Who Underwent PITA | Children Who Underwent T&A
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children Who Underwent PITA | Children Who Underwent T&A | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.33 (3.65) | 6.15 (3.29) | 5.74 (3.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 11
  Male | 12 | 7 | 19
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Apnea-hypopnea Index (AHI)
Description: Change in the number of apneas plus hypopneas per hour of sleep on preoperative sleep study compared to postoperative sleep study, Change is calculated as baseline minus 4-year time point
Time Frame: Baseline and 4 years
Measure: Median (Standard Deviation); unit: events per hour of sleep
Arm/Group | Children Who Underwent PITA | Children Who Underwent T&A
Number analyzed (Participants) | 15 | 15
events per hour of sleep | 3.8 (8.5) | 8.0 (18.7)
Statistical Analysis 1: Comparison: Children Who Underwent PITA vs Children Who Underwent T&A; The relationship of surgical group with AHI change was evaluated by constructing a mixed linear model (MLM). The dependent variable was the logarithm of the ratio of postoperative AHI score to preoperative AHI score; this transformation was chosen in order to minimize skew of model residuals. Surgical group was introduced as a fixed factor; subject pairs constituted levels of a random blocking) factor; Test type: Superiority or Other; p = .590, Mixed Models Analysis — A priori threshold for statistical significance was P<.05
Statistical Analysis 2: Comparison: Children Who Underwent PITA vs Children Who Underwent T&A; A mixed linear model was constructed as described above. Variance was estimated separately for each group; Test type: Superiority or Other; p = .022, Mixed Models Analysis — P value for the variances. The a priori threshold for statistical significance was P < .05

2. Secondary Outcome: Number of Patients With Apnea-hypopnea Index (AHI) Less Than or Equal to 5
Description: Number of patients with postoperative apnea-hypopnea index (apneas plus hypopneas per hour of sleep) less than or equal to 5 on sleep study
Time Frame: Baseline and 4 years
Measure: Number; unit: participants
Arm/Group | Children Who Underwent PITA | Children Who Underwent T&A
Number analyzed (Participants) | 15 | 15
participants | 5 | 4
Statistical Analysis 1: Comparison: Children Who Underwent PITA vs Children Who Underwent T&A; The relationship of surgical group with postoperative AHI ≤ 5 was evaluated by exact conditional logistic regression, predicting AHI ≤ 5 from surgical group with subject pairs as strata; Test type: Superiority or Other; p = 1.00, Fisher Exact

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Children Who Underwent PITA | Children Who Underwent T&A
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Selection bias, sample size limitation as it the study was not powered to detect small differences between the groups, and the use of unattended home PSG instead of laboratory-based PSG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No